CLINICAL TRIAL: NCT06403566
Title: THE EFFECT OF HAND AND BACK MASSAGE ON PAIN, SLEEP AND SELF-CARE IN WOMEN UNDERGOING HYSTERECTOMY: A RANDOMIZED CONTROLLED TRIAL
Brief Title: THE EFFECT OF HAND AND BACK MASSAGE ON PAIN, SLEEP AND SELF-CARE IN WOMEN UNDERGOING HYSTERECTOMY
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, seda karaçay yıkar, Assistant professor, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 139-43
Record Dates: First submitted 2024-05-03; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Sleep; Pain; Self Efficacy
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- hand massage application (Experimental): hand massage will be applied before and after surgery
  Interventions: Other: hand massage
- back massage application (Active Comparator): back massage will be applied before and after surgery
  Interventions: Other: hand massage
- control group (No Intervention): no intervention will be made

INTERVENTIONS:
Other: hand massage — three group randomized controlled trials
  Other Names: back massage
  Arms: back massage application; hand massage application

SUMMARY:
Postoperative incision pain is an acute pain that begins with the stimulation of neuroreceptors from surgical trauma and usually resolves within a few days. Today, the physiology of acute pain is better understood and new approaches to pain management are emerging. However, studies conducted in recent years have reported that postoperative pain management is inadequate, and therefore approximately 50-80% of patients still experience moderate to severe pain

DETAILED DESCRIPTION:
Self-care is the realization of health activities to maintain one's health, life and well-being (14). Self-care power is at different levels in each person and perceptual, cognitive, interpersonal and psychomotor characteristics are needed for an effective self-care power to be formed. Therefore, self-care power varies according to the ability and health status of the individual (12). According to Orem, the development and maintenance of health are the results to be obtained through self-care. Orem's theory also "values personal responsibility for health and indicates that nursing services may have a key role in prevention and health education". Since self-care is a learnable behavior, nurses can encourage and support people's self-care efforts and increase the individual's participation by providing health education (12).

When the literature is examined, there are a limited number of studies examining the effect of back massage on pain in women undergoing hysterectomy surgery. There are studies examining the effect of reiki on pain in different fields (13,14). Pain is a condition that affects all dimensions of the individual including biophysiologic, psychological, sociocultural and political-economic. Although analgesics are indispensable to alleviate postoperative pain, undesirable effects may occur when overused. Therefore, nurses' use of non-drug methods in addition to pharmacologic methods will increase the effectiveness of pharmacologic methods (15). Pharmacology

ELIGIBILITY:
Inclusion Criteria:

* Age range 25-65,
* Elective surgery,
* Lying in the hospital for at least 2 days after surgery,
* Operated under general anesthesia

Exclusion Criteria:

* No serious complications developed after surgery,
* Never had a back or hand massage before,
* Cognitive, effective and without any problem preventing communication,
* No psychiatric problems,
* Patients receiving a single type of analgesic drug (non-narcotic analgesics) to ensure homogeneity of the groups and to increase the reliability of the study results,
* Patients not using Patient Controlled Analgesia (PCA) will be included in the sample.

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — women undergoing hysterectomy surgery
Enrollment: 102 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
hand massage | will be checked on the 2nd postoperative day
  hand massage reduces women's pain score 0-10 points
back massage | will be checked on the 2nd postoperative day
  back massage women's pain score 76-100 points
hand massage | will be checked on the 2nd postoperative day
  hand massage improves women's scores by reducing sleep problems
back massage | will be checked on the 2nd postoperative day
  back massage improves women's scores by reducing sleep problems

CONTACTS AND LOCATIONS:
Locations (1):
- Seda Karaçay Yıkar, Adana, Sarıcam, Turkey (Türkiye)